CLINICAL TRIAL: NCT06678217
Title: Detection of Electrodermal Activity in Pain (DEEP)
Brief Title: Detection of Electrodermal Activity in Pain 1
Acronym: DEEP 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Kirstine Skov Benthien, Principal Investigator, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-24037808-Phase-1
Record Dates: First submitted 2024-11-01; First posted 2024-11-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Acute Pain
Keywords: pain; electrodermal activity; pain detection; pain prediction; galvanic skin response; wearable; pain monitoring
MeSH Terms: conditions — Acute Pain; Pain | interventions — Stroop Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPT only (Experimental): Participants go through the cold pressor test.
  Interventions: Other: Cold pressor test
- CPT and Stroop (Experimental): Participants go through the Stroop task before the cold pressor test.
  Interventions: Other: Stroop task; Other: Cold pressor test

INTERVENTIONS:
Other: Stroop task — The Stroop task will be used as a mild, acute stressor since it has effects on anxiety and autonomic response. In each Stroop task condition, four coloured visual stimuli will be presented on a computer screen for 3 s with 7 s inter-stimulus interval. The stimuli will be coloured words naming the colour of the ink in the nonconflict task condition (e.g. GREEN written in green ink) and a different colour in the conflict task condition (e.g. GREEN written in red ink). The participants were asked to name the colour of the stimuli. The test will be administered using the online version of PsyToolKit (Stoet, 2021).
  Arms: CPT and Stroop
Other: Cold pressor test — The participant lowers their hand in icy water to induce temporary tonic pain

SUMMARY:
The goal of this study is to investigate the association between self-reported pain and electrodermal activity and to develop an algorithm that detects pain-related changes in electrodermal activity in healthy volunteers undergoing a cold pressor test. The study is exploratory.

The main research questions are:

Can pain be detected using electrodermal activity, and do psychological variables, including stress, affect the electrodermal response to pain?

Study Design:

The study has two arms.

Methodology:

Thirty-seven healthy volunteers perform an experimental pain task while their electrodermal activity is recorded and complete questionnaires. The participants are randomized 1:1 to either the cold pressor test alone or the cold pressor test combined with a mild experimental stressor (Stroop task).

Analysis:

Discriminant analysis will be used to differentiate between mild, moderate, and severe pain levels. Secondary outcomes include assessing the influence of the mild stressor on the pain response. This study is exploratory, generating hypotheses for subsequent phases of the project.

DETAILED DESCRIPTION:
Methods Research Design The purpose of phase 1 is to develop an algorithm to assess and predict pain using biological signals and self-reported outcome measures. For phase 1, a randomized controlled trial design will be used. Group 1 will undergo the Cold Pressor Test (CPT) only, while Group 2 will undergo the CPT in addition to the Stroop task.

Measures Subjective measures (Self-Reported) Pain. Pain intensity (interval, 0 to 10) is measured using the numerical rating scale (NRS), a commonly used tool asking patients to rate their pain intensity on a scale from 0 to 10, with 0 indicating no pain and 10 reflecting the worst possible pain.

Pain Catastrophizing. It is measured using the Pain Catastrophizing Scale (PCS). This scale is short, and consists of 13-items scored on a 5-point Likert scale from 0 (not at all) to 4 (all the time).

Patient Health Status. The Patient Health Questionnaire is commonly used to provisionally diagnose depression and grade severity of symptoms in general medical and mental health settings. The PHQ-9 is the depression module.

Objective measures Electrodermal activity. A wearable device provided by Movisens GmbH will be used to record skin conductance measured in microsiemens (μS).

Cardiac activity. Additionally, 4-channel ECG signal with Texas Instruments ADS1299 will be used to collect data for calculating the periodic repolarization period (PRD).

Interventions & Apparatus

The Cold Pressor Test The CPT test will be used to induce tonic pain in phase 1.The CPT is a tonic pain stimulus where participants immerse their hand into 2 degrees Celcius cold water.

The Stroop task The Stroop task will be used as a mild, acute stressor.

Wearable device The EdaMove 4 device provided by Movisens GmbH consists of an EDA and activity sensor. It will be used to collect data during the entire experimental procedure including the CPT and Stroop task.

Texas Instruments ADS1299 amplifier Texas Instruments ADS1299 amplifier will be used to collect a 4-channel ECG signal to analyze the PRD during the tonic pain stimulation with the CPT.

Software Python, R and STATA will be used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Danish
* Age over 18

Exclusion Criteria:

* Presence of current pain
* Current use of analgesic medication
* Persistent or recurrent pain that exists for longer than 3 months
* Blood circulation or cardiovascular disorders
* Hypertension
* A skin condition on the to-be-tested body parts
* Raynaud syndrome
* Substance abuse
* Pregnancy or lactation and
* A current diagnosis with psychological/ psychiatric disorders
* Diagnosed with chronic illness
* Symptoms of an infectious disease
* PHQ-9 reveals suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | while participants have their wrist immersed in cold water for the Cold Pressor Test, for maximum 3 minutes.
  Numerical rating scale score. Pain intensity (interval, 0 to 10) is measured using the NRS, a commonly used tool asking patients to rate their pain intensity on a scale from 0 to 10, with 0 indicating no pain and 10 reflecting the worst possible pain.

SECONDARY OUTCOMES:
Skin conductance level | while participants wear the device throughout testing, which lasts up to fifteen minutes.
  The average skin conductance value (μS) for periods of 10 seconds.
Number of Skin Conductance Fluctuations | while participants wear the device throughout testing, which lasts up to fifteen minutes.
  Peaks with minimum amplitudes of 0.02 μS and a slope rate < 2 μS/s, in 10 second intervals.
Cold pressor endurance time | while participants have their wrist immersed in cold water for the Cold Pressor Test
  Maximum time of immersion in cold water.
The Patient Health Questionnaire (PHQ-9) | administered the day of testing
  The Patient Health Questionnaire (PHQ-9) will be used to screen participants as symptoms of depression in order to control during the statistical analysis.
  The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day), providing a 0 to 27 severity score.
Pain Catastrophizing | administered the day of testing
  It is measured using the Pain Catastrophizing Scale (PCS). This scale is short, and consists of 13-items scored on a 5-point Likert scale from 0 (not at all) to 4 (all the time), asking participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain
  Higher scores indicate higher levels of pain catastrophizing and the total score range varies from 0 to 52.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine Skov Benthien, PhD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital - Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No